CLINICAL TRIAL: NCT03468517
Title: Does the Preoperative Anxiety Decrease With BATHE Method? A Prospective Randomized Study
Brief Title: Preoperative Anxiety and BATHE Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Derya Arslan Yurtlu, Associate Professor Dr, MD, Izmir Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KÇÜ-IATRH
Record Dates: First submitted 2017-12-11; First posted 2018-03-16 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Anxiety State
Keywords: General Anaesthesia; Preoperative Anxiety; BATHE method
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Standard preoperative evaluation process will continue without any intervention.
- Bathe Group (Active Comparator): In the comparator group of patients, Bathe method will be applied at preoperative evaluation process.
  Interventions: Other: Bathe method:

INTERVENTIONS:
Other: Bathe method: — BATHE technique, on the other hand, is one of the short therapeutic consultation techniques that strengthen the doctor-patient relationship. BATHE stands for the initials of the questions that include the titles for Background, Affect, Trouble, Handling and Empathy. It allows evaluating the physiological stress of the patients quickly. BATHE method necessitates an empathetic expression that includes the view of the patient in addition to asking the key questions by the doctor doing the interview
  Arms: Bathe Group

SUMMARY:
The patients were randomized into "Bathe" and "Control" groups by using the closed envelope technique. Demographic data and pre-examination anxiety scores State- Trait Anxiety Inventory (STAI) are recorded as entrance STAI for all patients. Then they had routine preoperative evaluation. During these procedures, Bathe method was applied to the Bathe Group whereas it was not applied to the Control Group. After that post-examination, STAI scores were recorded as exit STAI and the patients were later asked questions about their contentment.

DETAILED DESCRIPTION:
Participants and Procedure:

Before the study, approval from the ethics committee of Katip Celebi University Faculty of Medicine was received. 463 patients were included in the prospective randomized double blind study. To accept to be involved in the study, being above 18 years old and being literate were the criteria necessary to be involved in the study. Exclusion criteria were listed as below: Not to accept to be involved in the study, being under 18 years old, being illiterate, having been diagnosed a psychiatric illness, having a physical/psychiatric trauma within the last one year, using sedative, antidepressant, antiepileptic substances or drugs, having cooperation, understanding or hearing problems, belonging to American Society of Anesthesiologists (ASA) physical situation (PS) III and above.

STAI Analysis:

By randomization using the closed envelope technique, the envelopes have been prepared beforehand the patient examination. Sealed envelopes contained a specific number and a patient group defined for this number. Thus, patients were divided into two as 'bathe group' and 'control group' by simple randomization method and they were given one of these closed envelopes respectively.

The demographic data of the patients which included their names-surnames, gender, age, educational background, income level, their previous anesthesia experience (no experience, with general anesthesia experience, with regional anesthesia experience, with both general and regional anesthesia experience) have been questioned. Following this, STAI anxiety questionnaire that was validated to Turkish language by Oner et al., has been applied in order to learn the patients' anxiety levels before preoperative evaluation and the result has been recorded as entrance STAI. Since we aimed to decrease operation anxiety of the patients, we only used state anxiety scale at that moment. After then, patients have been taken to anesthesia examination room.

BATHE technique:

All the patients were evaluated before the anaesthesia. Later, by opening the envelope of the patient, his/her group has been learned. Feedback has been given with empathetic statements to those in BATHE group after key questions and they have been informed about the possible outcomes . Bathe questions have been modelled by Hepner et al. and have been modified in order to be used in perioperative period. It was validated to Turkish language by Akturan et al. For the patients in the control group, the interview ended by routine preoperative evaluation (without applying BATHE technique).

Satisfaction Questionnaire At the end of the examination, the STAI anxiety questionnaire (Exit STAI) was repeated for patients to measure their anxiety levels. In addition, satisfaction questionnaire, which was prepared by Leiblum et al., was also applied. Patients have been asked to rate their satisfaction level by using five point Likert scale.

At the end, the bathe method has also been applied to the patients in control group as well. The reason for this procedure was to prevent the discrimination of the control group. Obviously, this did not change the results of the study as the satisfaction questionnaire was applied before the BATHE technique procedure for the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old

Exclusion Criteria:

* Not to accept to be involved in the study
* Being illiterate
* Having been diagnosed a psychiatric illness
* Having a physical/psychiatric trauma within the last one year
* Using sedative, antidepressant, antiepileptic substances or drugs
* Having cooperation, understanding or hearing problems
* Patients who were ASA PS >III

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-03-30 (Actual)

PRIMARY OUTCOMES:
2 item State Trait Anxiety Intentory (STAI) Score Measure | 1 hour
  State Trait Anxiety Intentory (STAI) Score Measure was applied before BATHE intervention. Then, State Trait Anxiety Intentory (STAI) Score Measure was again applied after BATHE intervention. Then, the change between STAI scores are assessed to understand whether BATHE intervention makes a difference or not.

SECONDARY OUTCOMES:
Patient satisfaction score | 1 hour
  Five point Likert scale were applied to determine patient satisfaction after preoperative anesthesia evaluation. Patient satisfaction is scored 11-55. (11=no satisfaction, 55=much satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Pınar P Ayvat, MD, Study Chair — Principal Investigator; Derya DA Yurtlu, MD, Principal Investigator — Investigator; Yasemin Y Işık, MD, Principal Investigator — Investigator; Uğur U Özgürbüz, MD, Principal Investigator — Investigator; Fatma F Güntürkün, PhD, Principal Investigator — Investigator; Kaan K Katırcıoğlu, MD, Principal Investigator — Investigator; Mehmet M Kızılkaya, MD, Principal Investigator — Investigator
Locations (1):
- Katip Çelebi University İzmir Atatürk Training and Reseach Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leiblum SR, Schnall E, Seehuus M, DeMaria A. To BATHE or not to BATHE: patient satisfaction with visits to their family physician. Fam Med. 2008 Jun;40(6):407-11. PMID 18773778

DOCUMENTS (1):
  • Study Protocol (2015-11-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT03468517/Prot_000.pdf